CLINICAL TRIAL: NCT06256094
Title: The Effects of a2 Infant Formula on Growth and Tolerance in Healthy Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: a2 Milk Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A2220616005
Record Dates: First submitted 2024-01-15; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a2 Platinum Premium Infant Formula Stage 1 (Experimental): a2 Platinum Premium Stage 1 (0-6 months) cow's milk based powder infant formula
  Interventions: Dietary Supplement: a2 Platinum Premium Infant Formula Stage 1
- Frisolac Infant Formula Stage 1 (Dutch Edition) (Active Comparator): Dutch Edition of the Frisolac Stage 1 (0-6 months) cow's milk based powder infant formula
  Interventions: Dietary Supplement: Frisolac Infant Formula Stage 1 (Dutch Edition)

INTERVENTIONS:
Dietary Supplement: a2 Platinum Premium Infant Formula Stage 1 — Oral intake of a2 Platinum Premium Infant Formula Stage 1 milk powder (dissolved in water)
  Arms: a2 Platinum Premium Infant Formula Stage 1
Dietary Supplement: Frisolac Infant Formula Stage 1 (Dutch Edition) — Oral intake of Frisolac Infant Formula Step 1 (Dutch Edition) milk power (dissolved in water)
  Arms: Frisolac Infant Formula Stage 1 (Dutch Edition)

SUMMARY:
This is a randomized, open-label, prospective study to evaluate the nutritive effects of an a2 infant formula on growth and tolerance in healthy term infants. A total of 280 healthy, term, mixed-fed infants between 60 and 120 days of age were enrolled at Shanghai. The participants were randomly assigned to one of the two study groups: the a2 infant formula group and the conventional A1/A2 infant formula group. Each group contained 140 infants. The study duration was 56 days.

DETAILED DESCRIPTION:
Primary objective:

To compare the growth measurements of the infants fed with the a2 infant formula with those fed with conventional A1/A2 infant formula during the study period.

Secondary objectives:

To compare the two study groups in

1. Dermatitis quality of life
2. Formula tolerability and acceptability
3. All medically confirmed adverse events

The study included four visits at day 0 (baseline), day 14, day 28 and day 56. Information of efficacy outcomes were collected at each visit. Subject diary was used to record tolerance data and daily formula feeding amount during the study. The parents of the participants were also required evaluate their satisfaction with the study formula at the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and term infants (37-42 weeks gestation);
* Birth weight between 2500g and 4500g;
* 60-120 days of age after birth;
* Mixed-fed: Infants who were fed with a mixture of formula and human milk, and received daily formula consumption of more than 400ml;
* Signed informed consent obtained form the guardian(s) of the infants;
* Parent or guardian of infant agrees not to enroll infant in another interventional clinical research survey while participating in this survey.

Exclusion Criteria:

* Congenital anomaly or hereditary/chronic/congenital diseases that could interfere with the study product evaluations;
* Evidence of feeding difficulties or intolerance/allergy to cow's milk;
* Conditions requiring infant feedings other than those specified in the protocol;
* Significant systemic disorders (cardiac, respiratory, endocrinological, hematologic, gastrointestinal, or other) or parental refusal to participate;
* Acute infection or gastroenteritis at the time of enrollment;
* Participation in other clinical trials at the time of the study;
* Investigator's uncertainty about the willingness or ability of the parents to comply with the protocol requirements.

Ages: 60 Days to 120 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Body weight measured in gram. | Baseline, Day 14, Day 28, Day 56
  Body weight measured in gram.

SECONDARY OUTCOMES:
Body length measured in centimeter. | Baseline, Day 14, Day 28, Day 56
  Body length measured in centimeter.
Head circumference measured in centimeter. | Baseline, Day 14, Day 28, Day 56
  Head circumference measured in centimeter.
Body mass index calculated from body weight and length. | Baseline, Day 14, Day 28, Day 56
  Body mass index calculated from as weight (kg) dived by the square of body length (meter).
Weight-for-age Z-score that describe the distance and direction of the weight of a participant away from the mean of the population of the same age | Baseline, Day 14, Day 28, Day 56
  A standard score for measuring weight growth calculated according to the WHO Growth Standards. The weight-for-age Z-score is the distance and direction of the weight of a participant away from the mean body weight of the population of the same age.
Length-for-age Z-score that describe the distance and direction of the body length of a participant away from the mean body length of the population of the same age | Baseline, Day 14, Day 28, Day 56
  A standard score for measuring body length growth calculated according to the WHO Growth Standards. The length-for-age Z-score is the distance and direction of the body length of a participant away from the mean body length of the population of the same age.
BMI-for-age Z-score that describe the distance and direction of the body mass index of a participant away from the mean body mass index of the population of the same age | Baseline, Day 14, Day 28, Day 56
  A standard score for measuring body mass index (BMI) calculated according to the WHO Growth Standards. The BMI-for-age Z-score is the distance and direction of the body mass index of a participant away from the mean body mass index of the population of the same age.
Head circumference-for-age Z-score that describe the distance and direction of the head circumference of a participant away from the mean head circumference of the population of the same age | Baseline, Day 14, Day 28, Day 56
  A standard score for measuring head circumference calculated according to the WHO Growth Standards. The head circumference-for-age Z-score is the distance and direction of the head circumference of a participant away from the mean head circumference of the population of the same age.
Weight-for-length Z-score that describe the distance and direction of the weight of a participant away from the mean weight of the population of the same body length | Baseline, Day 14, Day 28, Day 56
  A standard score for measuring weight-for-length growth calculated according to the WHO Growth Standards. The weight-for-length Z-score is the distance and direction of the body weight of a participant away from the mean body weight of the population of the same body length.
Infants' gastrointestinal symptom score evaluated using the Infant Gastrointestinal Symptom Questionnaire (IGSQ) | Baseline, Day 14, Day 28, Day 56
  The IGSQ score is the sum of 5 domains scores of stooling, spitting up/vomiting, crying, fussiness and flatulence, derived by summing up the relating raw individual scores. Each raw score range from 0 to 5, with higher score indicating more severe gastrointestinal symptoms. Data was collected daily, and the average score during the past week of each visit was used for analyses.
Number of crying periods evaluated in each 15-minutes period during a day | Baseline, Day 14, Day 28, Day 56
  Number of 15-minute periods at morning, afternoon, evening and night, and the daily total number of crying periods. Data was collected daily, and the average daily number of crying periods during the past week of each visit was used for analyses.
Infants' Dermatitis Quality of Life Index (IDQoL) that measured participants' quality of life related to dermatitis | Baseline, Day 14, Day 28, Day 56
  An index to evaluate the quality of life related to dermatitis during the past week of each visit. The IDQoL index is the sum of one score for evaluating dermatitis severity (range from 0 to 4 indicating increasing severity from no symptom to very servere symptom) and 10 individual scores (each range from 0 to 3 indicating increasing frequency from none to very often) evaluating the possible problems encountered in daily life due to dermatitis, including itching and scratching, mood, time to get to sleep, sleep disturbance, disturbed playing or swimming, disturbed family activities, problems during meal times, problems from treatment, problems at dressing, and problems at bath time.
Average daily formula intake amount (ml/day) during the past week measured by formula intake diary | Baseline, Day 14, Day 28, Day 56
  Daily formula intake amount was recorded in ml. The average daily formula intake amount during the past week of each visit was used to assess formula feeding amount.
Percent of participants with relieved gastrointestinal symptoms by the end of the study, evaluated using the Formula Satisfaction Questionnaire | Day 56
  Parents were required to report whether the gastrointestinal symptoms of the participant have been relieved by the end of the study. Dichotomized variable with 2 levels: Yes or No.
Percent of participants with relieved skin symptoms by the end of the study, evaluated using the Formula Satisfaction Questionnaire | Day 56
  Parents were required to report whether participant's skin symptoms such as eczema or dermatitis have been relieved by the end of the study. Dichotomized variable with 2 levels: Yes or No.
Percent of parents of the participants with intention of continuing to feed the child with the study formula, measured in 3 levels: Yes, No, or Not sure using the Formula Satisfaction Questionnaire | Day 56
  Parents were required to indicate their intention of continuing to feed the child with the study formula. Categorical variable with 3 levels: Yes, No, or Not sure.
Percent of overall satisfaction levels with the study formula, measured in 4 levels: Satisfied, Neutral, Dissatisfied, or Not sure using the Formula Satisfaction Questionnaire | Day 56
  Overall satisfaction with study formula was evaluated by the parents at the end of the study. Category variable with 4 levels: Satisfied, Neutral, Dissatisfied, or Not sure.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Wang, Study Director — Adjuvant Advertising (Shanghai) Co., Ltd
Locations (1):
- Shanghai Weierkang Pediatric Outpatient Department, Shanghai, China

REFERENCES:
- [Derived] Li J, Yang T, Sheng X. Effect of Infant Formula Made With Milk Free of A1-Type beta-Casein on Growth and Comfort: A Randomized Controlled Trial. Food Sci Nutr. 2025 Jul 15;13(7):e70606. doi: 10.1002/fsn3.70606. eCollection 2025 Jul. PMID 40672544